CLINICAL TRIAL: NCT00144287
Title: An Open Label Safety Study of Tipranavir Co-Administered With Low-Dose Ritonavir (TVP/r) in Patients With Advanced HIV-1 Infection and Limited Treatment Options
Brief Title: Safety Study of Tipranavir Co-administered With Low-dose Ritonavir (TPV/r) in Patients With Advanced HIV-1 Infection and Limited Treatment Options
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.68
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir

INTERVENTIONS:
Drug: Tipranavir/Ritonavir

SUMMARY:
This study evaluated the safety and tolerability of tipranavir to improve treatment options for HIV type 1-infected patients who have been previously treated and whose treatment is no longer effective.

DETAILED DESCRIPTION:
The purpose of this open label study is to assess the safety and tolerability of tipranavir co-administered with low-dose ritonavir (500 mg tipranavir/200 mg ritonavir BID) in HIV-1 infected patients who are triple antiretroviral class experienced with at least two previous PI-containing regimens.

The safety assessment will be performed by evaluating:

* The frequency of treatment-emergent adverse events (AEs) , all serious adverse events (SAEs), and additional safety laboratory parameters.
* The occurrence of PI class-specific AEs, such as hemorrhage, dyslipidemia, hepatic events, hyperglycemia, pancreatitis, and rash.

The efficacy assessment will be performed by evaluating:

* The quantity of HIV-1 RNA
* The CD4 cell count.

Study Hypothesis:

The purpose of this open label study is to assess the safety and tolerability of tipranavir co-administered with low-dose ritonavir (500 mg tipranavir/200 mg ritonavir BID) in HIV-1 infected patients who are triple antiretroviral class experienced with at least two previous PI-containing regimens.

Comparison(s):

N.A.

ELIGIBILITY:
Inclusion Criteria:

1. Triple antiretroviral class experienced patients with at least two previous PI-based regimens, who had failed or are intolerant to currently approved HIV-1 treatments
2. Age >= 18 years
3. Patient is willing to use an effective barrier method of contraception for the duration of study participation and up to three months thereafter
4. Patient voluntarily provides written informed consent to participate, in compliance with local law

Exclusion Criteria:

1. Hypersensitivity to active ingredients or any of the excipients in tipranavir or ritonavir
2. Required use of restricted medications
3. Female patients of childbearing potential who:

   * Have a positive pregnancy test at baseline or
   * Are breast feeding.
4. Any medical condition(s) which, in the opinion of the investigator, would interfere with the patient´s ability to participate in or adhere to the requirements of this protocol.
5. Use of other investigational drugs, within 30 days prior to TPV/r initiation and for the duration of study participation.
6. Hepatic impairment(*) evidenced by the following baseline laboratory findings:

   * AST or ALT >5X upper limit of normal (ULN) or total bilirubin >3.5X ULN or
   * AST or ALT >2.5X ULN and total bilirubin >2X ULN

(*) Patients with liver enzymes outside this range will be restricted from participation in this safety study until more data become available from ongoing phase III clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2004-05; Primary Completion 2006-04 (Actual); Study Completion 2006-04

PRIMARY OUTCOMES:
The frequency of treatment-emergent adverse events (AEs), all serious AEs, and additional safety laboratory parameters
The occurrence of PI class-specific AEs, such as hemorrhage, dyslipidemia, hepatic events, hyperglycemia, pancreatitis, and rash

SECONDARY OUTCOMES:
The quantity of HIV-1 RNA
The CD4 cell count

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (40):
- Germany (40):
  - Boehringer Ingelheim Investigational Site, Aachen
  - Boehringer Ingelheim Investigational Site, Berlin
  - Epimed GmbH, Berlin
  - Universitätskliniken Charité, Berlin
  - Klinikum der Ruhr-Universität Bochum, Bochum
  - Medizinische Universitätsklinik Bonn, Bonn
  - Krankenhaus der, Cologne
  - Boehringer Ingelheim Investigational Site, Cologne
  - Universitätsklinik Köln, Cologne
  - Klinikum Dortmund g GmbH, Dortmund
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Boehringer Ingelheim Investigational Site, Duisburg
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Boehringer Ingelheim Investigational Site, Düsseldorf
  - Universitätsklinik Erlangen-Nürnberg, Erlangen
  - Universitätsklinikum Essen, Essen
  - Klinikum der J.-W.-Goethe-Universität, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - Klinikum der Justus-Liebig-Universität, Giessen
  - ifi Institut für Interdisziplinäre Infektiologie, Hamburg
  - IPM Study Center GmbH, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Boehringer Ingelheim Investigational Site, Hanover
  - Med. Hochschule Hannover, Hanover
  - Universitätsklinik des Saarlandes, Homburg/Saar
  - Universitätsklinikum im, Kiel
  - Städtisches Krankenhaus Kemperhof, Koblenz
  - Städtisches Klinikum St. Georg, Leipzig
  - Johannes-Gutenberg-Universität Mainz, Mainz
  - Boehringer Ingelheim Investigational Site, München
  - Medizinische Poliklinik, München
  - Boehringer Ingelheim Investigational Site, Münster
  - Klinik und Poliklinik für Neurologie, Münster
  - Boehringer Ingelheim Investigational Site, Nuremberg
  - Boehringer Ingelheim Investigational Site, Oldenburg
  - Klinium Natruper Holz, Osnabrück
  - Klinikum Salzgitter GmbH, Salzgitter
  - Boehringer Ingelheim Investigational Site, Stuttgart
  - Medizinische Universitätsklinik Ulm, Ulm
  - Boehringer Ingelheim Investigational Site, Wuppertal